CLINICAL TRIAL: NCT04704778
Title: Randomized Clinical Trial of Electrostimulation Therapies With Implementation of Multifractal Electromyographic Analysis for Patients With Temporomandibular Disorders
Brief Title: Electrostimulation Therapies With Implementation of Multifractal Electromyographic Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Universidad de la Republica (Other); Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government); Centro De Investigación Y De Estudios Avanzados Del Instituto Politécnico Nacional-Unidad Irapuato (Other); Facultad de Estudios Superiores Iztacala, UNAM. (Unknown)
Responsible Party: Principal Investigator, Claudia Ivonne Rodriguez Castañeda, Master of Clinical Dental Sciences, Universidad Nacional Autonoma de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIE/0508/02/2020
Record Dates: First submitted 2020-12-15; First posted 2021-01-12 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Temporomandibular Dysfunction (TMD); Orofacial Pain
Keywords: Electromyographic; Electrostimulation therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Facial Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The selected sample will be divided into three groups (GA = transcutaneous electrostimulation and splint, GB = percutaneous electrostimulation and splint, GC = splint); the allocation by group will be made by means of a randomization in balanced blocks. For this process, a series of blocks will be assembled made up of a certain number of cells in which the types of treatment are included. The number of blocks will be determined by the number of participants to be included in the study and the number of cells that it has been decided to include in each block. Each block will contain in each cell one of the treatment alternatives and within each block there must be a balanced number of possible treatments.
Who Masked: Outcomes Assessor
Masking Description: Blind observer:
  A third party (statesman) is used, who does not know the treatment that each person is receiving.
  patient, to assess the response.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Transcutaneous (Active Comparator): Transcutaneous electrostimulation and uso of oclusal splint
  Interventions: Combination Product: Transcutaneus electrostimulation therapies; Combination Product: Percutaneus electrostimulation therapies; Diagnostic Test: Oclusal splint
- Percutaneous (Active Comparator): Percutaneous electrostimulation and splint
  Interventions: Combination Product: Transcutaneus electrostimulation therapies; Combination Product: Percutaneus electrostimulation therapies; Diagnostic Test: Oclusal splint
- Control (Placebo Comparator): Oclusal splint
  Interventions: Diagnostic Test: Oclusal splint

INTERVENTIONS:
Combination Product: Transcutaneus electrostimulation therapies — Sterile steel acupuncture needles of 0.25x13mm, disposable AcuBEST brand, and portable electro-stimulator equipment KWD- will be used. The superficial area of the skin of the masseter muscle will be cleaned with alcohol.
  Two needles will be placed in each masseter muscle, the area to be punctured is the origin of the masseter muscle or superficial area of the mandibular condyle anterior to the atrial tragus approximately 1cm away, insertion of the masseter muscle at the angle of the mandible. The two double alligator cables will be connected to the head of the needles. The positive pole will be connected at the origin of the masseter muscle and the negative pole at the insertion.
  The parameters to be used will be are two frequency bands (210Hz-10140Hz.); amplitude 3050 volts, pulse duration: 40100 msec; and the output intensity: 0.70 (for 100Hz). The treatment time will be 20 minutes.
  Other Names: Electroacupuntur
  Arms: Percutaneous; Transcutaneous
Combination Product: Percutaneus electrostimulation therapies — Kendall® MediTrace 100 conductive adhesive ECG electrodes (pediatric) 2.4 cm in diameter, and portable KWD-808 electrostimulator equipment will be used.
  The superficial area of the skin will be cleaned, two electrodes will be placed on each muscle (superficial area of the mandibular condyle and at the angle of the jaw). The current leads will then be connected to the KWD-808 electroacupuncturist to the patient.
  Current will be transmitted with a square waveform, 210Hz-10140Hz of frequency, 3050 volts of amplitude and 40100 msec pulse time. The treatment time will be 20 minutes.
  Other Names: TENS
  Arms: Percutaneous; Transcutaneous
Diagnostic Test: Oclusal splint — The occlusal splint is worn 24 hours a day, removed for eating and brushing teeth. It is washed with neutral liquid hand soap.
  For the preparation, an impression of the maxillary dental arches will be taken with alginate; It is made with acetate .060 and .080.
  Relining is done with self-curing acrylic on the occlusal surface of the splint
  Other Names: Control

SUMMARY:
The objective is to compare the neuromuscular electrical activity and muscle fatigue of the masseter muscles in three groups of patients with different treatments for TMD (GA = Transcutaneous electrostimulation and splint, GB = percutaneous electrostimulation and splint, and GC = Occlusal splint) by means of 6 electromyographic recordings scheduled weekly.

The study population will be patients with TMD who will enter the Physiology Laboratory of the Division of Postgraduate Studies and Research (DEPeI) UNAM, admitted during the period from March to December 2021 The selection of the sample will be carried out by convenience sampling which will be carried out based on the clinical evaluation (considering the inclusion and exclusion criteria). The recruitment period will take place during the period from March to December 2021.

The selected sample will be divided into three groups (GA = transcutaneous electrostimulation and splint, GB = percutaneous electrostimulation and splint, GC = splint); the allocation by group will be made by means of a randomization in balanced blocks. The total sample size calculated for this study was 84 patients, 28 for each group.

The diagnostic process of Temporomandibular Dysfunction (TMD) will be carried out by the Principal Investigator using the Diagnostic Criteria and Investigation of Temporomandibular Disorders (CDI / TMD).

DETAILED DESCRIPTION:
Temporomandibular dysfunction or disorder (TMD) is a functional disorder of the temporomandibular joint (TMJ), and is the cause of non-dental pain in the orofacial region.

TMD presents diagnostic difficulties, the literature suggests objective assessment of neuromuscular activity. Electromyography (EMG) is a reliable tool to determine the degree of functional muscle alteration, the EMG signal can be estimated and characterized by multifractal analysis, for example, the Hurts Index. This method is used successfully in the study of physiological signals with high biological variability (signals: cardiac, cardiovascular, ophthalmological, neuronal, metabolic, etc.), it is considered suitable for the comprehensive analysis of neuromuscular behavior.

The objective is to compare the neuromuscular electrical activity (RMS) and muscle fatigue (Hurst index) of the masseter muscles in three groups of patients with different treatments for TMD (GA = Transcutaneous electrostimulation and splint, GB = percutaneous electrostimulation and splint, and GC = Occlusal splint) by means of 6 electromyographic recordings scheduled weekly.

The clinical examination will be performed in the order of the hands of the clock, beginning with the upper right quadrant. The first review will correspond to the presence of mixed dentition, use of prostheses, number of teeth, muscle pain (with a pressure algometer applying 1.5 kg / cm2 in masseter muscles, and 2.4 kg / cm2 in temporal muscles), joint pain (with algometer pressure applying 1.5 kg / cm2), presence of noises, limitation to mouth opening (with Terabite) and heart rate.

To assess pain by means of muscle and joint palpation with an algometer, the patient will be seated in a relaxed position, the evaluator will place the fine circular surface of the algometer perpendicular to the skin and an increasing pressure of 0.5 kg / cm2 will be applied increasing gradually over one minute until reaching 1.5 kg / cm2.

The patient will be instructed to verbalize the moment when pressure was exerted if a painful sensation was caused by muscle and in the joint area.

Treatment for TMD will be carried out using conventional treatment with an occlusal splint and as an auxiliary method, transcutaneous and percutaneous electrostimulation therapies will be applied by the same operator. The clinical control appointments for signs and symptoms of TMD, splint fitting, electromyographic records and application of electrostimulation therapy as an adjunct to the use of splint, will be scheduled once a week in the Physiology Laboratory during the hours of 9:00 a.m. 1:00 pm and 2:00 pm to 6:00 pm for six consecutive weeks.

The electromyographic recording technique was standardized (Cohen's Kappa 0.7). The recording system (hardware and software) that will be used for the electromyographic evaluation is the Electromyograph 1.2 UNAM-CINVESTAV, which consists of a two-channel system for the analysis of the electromyographic signal that offers greater precision and facilitates muscle assessment through the estimation made by the software of the RMS for its acronym in English (Root Mean Square) and Hurts Index.

The RMS and Hurts Index will be recorded using three electrodes: one placed at the muscular origin, another at the insertion, and finally one in the behind-the-ear area as a ground or neutral electrode. The RMS recording is performed at maximum intercuspation for 30 seconds; the action potential that is expressed in electrical energy will be recorded in microvolts per second (μV / s).

6 electromyographic recordings will be performed on each patient (one record each week) during the time of splint use. Electromyographic recordings will be scheduled as well as follow-up control appointments, to make adjustments to the physiological occlusal splint.

The transcutaneous electrostimulation therapy will be carried out by the Principal Investigator, who will be trained in the ISSSTE Clínica de Especialidades Oriente Leonardo Bravo Complex in the acupuncture service under the guidance of Dr. Roberto Sánchez Ahedo. (Surgeon, Specialist in Family Medicine. Training in acupuncture in different institutions. Master in Medical Education, Doctorate in Education, Professor of various courses in acupuncture from a medical perspective. Academic of the Faculty of Medicine of UNAM.) It will be completed the training process for the application of electrostimulation therapies based on the WHO Guidelines established in the Official Mexican NOM-172-SSA1-1998, which specifies the operating criteria for the practice of human acupuncture and related methods (electrostimulation therapies). The Standard governs that the training of a Physician or Health Personnel to fully exercise these therapies requires training of at least 350 academic hours. For this reason, the principal investigator will complete during this stage the theoretical, practical and clinical preparation course taught by the UNAM Faculty of Medicine "Diploma in Complementary Medicine and Acupuncture" with a total of 450 academic hours lasting one year (August 2019-February 2021), to comply with the training guidelines and basic training for the application of electrostimulation therapies.

For transcutaneous electrostimulation therapy, Kendall® MediTrace 100 conductive adhesive ECG electrodes (pediatric) with a diameter of 2.4 cm, and portable electro-stimulator equipment KWD-808 (professional equipment for electroacupuncture and rehabilitation) will be used.

The patient will be positioned in the dental chair, the superficial area of the skin of the masseter muscle will be cleaned with alcohol and cotton. Two Kendall® MediTrace 100 electrodes will be placed in each masseter muscle (right and left), considering the same references that were used for the electrodes placed for the electromyographic recording; the first electrode is placed at the origin of the masseter muscle or superficial area of the mandibular condyle and the second at the insertion of the masseter muscle at the angle of the mandible. After placing the electrodes, the KWD-808 electroacupuncture device will be connected to the patient by means of two double alligator cables; the alligators will be pressed to the metal head of each electrode: the positive pole (red color) will be connected at the origin of the masseter muscle and the negative pole (black color) at the insertion of the masseter muscle.

Before nerve stimulation, all patients will be informed of the perceived sensation, which in some patients will range from imperceptible to barely noticeable or not very noticeable.

The parameters to be used will be: pulse duration until sensory activation and high intensities, but with an established limit to prevent muscle contraction and that allows maximum comfort for 20 minutes. Current will be transmitted with square or rectangular waveform, the stimulation frequency: two frequency bands (low: 210Hz and high 10140Hz.); wave amplitude: 3050 volts, pulse duration: 40100 msec; and the output intensity: 0.70 (for 100Hz). The treatment time will be 20 minutes; the equipment has the quality of timing itself and after time it will stop transmitting a signal to the patient. The treatment will consist of the application of six consecutive therapies programs weekly.

The transcutaneous electrostimulation therapy will be carried out by the Principal Investigator, who will be trained in the ISSSTE Clínica de Especialidades Oriente Leonardo Bravo Complex in the acupuncture service under the guidance of Dr. Roberto Sánchez Ahedo.

Sterile steel acupuncture needles of 0.25x13mm, disposable AcuBEST brand (FDA 510K), and portable electrostimulator equipment KWD-808 (professional equipment for electroacupuncture and rehabilitation) will be used for percutaneous electrostimulation therapies.

Prior to the placement of therapy, the superficial area of the skin of the masseter muscle will be cleaned with alcohol and cotton. The puncture technique will be carried out by taking the needle through the body (not by the handle), the lower part is held between the thumb and index finger of the right hand, allowing the tip of the needle to pass. Directing the needle to the acupuncture point to insert it quickly (penetrating 5 mm).

Two needles will be placed in the right masseter muscle and two in the left masseter muscle, each one at the reference trigger points (local TMD points), following the "Practical recommendations for the treatment of Temporomandibular Disorders"; the area to be punctured is the origin of the masseter muscle or superficial area of the mandibular condyle anterior to the atrial tragus approximately 1cm away (proximal acupuncture points: Gb3, Si 19, Gb 2, St 7), insertion of the masseter muscle at the angle of the mandible (Proximal acupuncture points: St6, St5). For this study, distal stitches will not be placed.

After placing the needles, the KWD-808 electroacupuncture device will be connected to the patient; The two double alligator cables will be connected to each patient by means of the alligators that will directly press the head of the needles. The positive pole (red color) will be connected at the origin of the masseter muscle and the negative pole (black color) will be placed at the insertion of the masseter muscle.

Before nerve stimulation, all patients will be informed of the perceived sensation, which in some patients will range from imperceptible to barely noticeable or not very noticeable.

The treatment will be carried out every week with a total of six continuous therapies or if the patient deserves it until the remission of symptoms.

The recruitment phase of the sample will be carried out by evaluating the patients, the TMD diagnostic process and the evaluation of inclusion criteria that attend the Physiology Laboratory of DEPeI UNAM during the period from August to December 2020. The randomization will be carried out of patients recruited during this period.

The clinical methodology for the application of the therapies Transcutaneous electrical nerve stimulation and Percutaneous Neuromodulation Therapy will be carried out based on:

* OFFICIAL MEXICAN STANDARD NOM-017-SSA3-2012. Regulation of health services for the practice of human acupuncture and related methods.
* Official Mexican STANDARD NOM-197-SSA1-2000. That establishes the minimum infrastructure and equipment requirements for hospitals and specialized medical care offices.

ELIGIBILITY:
Inclusion Criteria:

* Patients assigned to the DEPeI Physiology Laboratory.
* Age range 18 to 60 years
* Without prior treatment of TTM or DTM
* Permanent dentition
* With malocclusion
* With prosthetic or implant treatments
* Partially toothless arches
* Bruxists
* Deviation to mandibular opening or closure
* Presence of joint noises depending
* Myofascial or joint pain

Exclusion Criteria:

* Degenerative joint disease
* Periodontal problems
* Orthodontic treatment
* Apparent neurological or sensory disabilities
* Patients with bleeding disorders or with anticoagulant intake
* Patients with pacemakers, defibrillators, or heart conditions
* Epilepsy, thrombophlebitis, active or uncontrolled phlebitis
* Facial wounds or severe acne
* Apparent Neurological or muscular disorders
* Allergic to metal
* Acute inflammatory processes or infections
* Pregnant
* Joint surgical history
* Malignancies
* Degenerative bone diseases
* Fibromyalgia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular electrical activity | Two months (every week with a total of six continuous records)
  Mathematical Root Mean Square (RMS) value Micro Voltios (µV.) determined by the EMG UNAM-CINVESTAV program, which represents the average of the squared values of the electromyographic activity of the right and left masseter muscles.
Muscular fatigue | Two months (every week with a total of six continuous records)
  Micro Voltios (µV.) Mathematical Hurst Index value determined by the EMG UNAM-CINVESTAV program, which represents the average of the squared values of the electromyographic activity of the right and left masseter muscles

SECONDARY OUTCOMES:
Temporomandibular dysfunction (DTM) | Day 1
  Functional alteration of the temporomandibular joint that is identified by the presence of muscle or joint pain, joint sounds and restriction, deviation or deflection in the mandibular opening.
  Patients diagnosed with DTM by CDI / TTM
Muscle pain | Two months (every week with a total of six continuous records)
  Amount of muscular pain reported by the patient when applying a pressure of 1.5 Kg / cm2 in masseter muscles and 2.4 Kg / cm2 in temporal muscles using a circular tip of a Baseline brand pressure algometer.Where 0 represents the absence of perceived pain, and 10 the maximum amount of pain
Limitation of mouth opening | Two months (every week with a total of six continuous records)
  Amount of millimeters measured from the incisal edge of the upper anterior teeth to the incisal edge of the lower anterior teeth with a TeraBite ruler. Opening limitation (<40mm.)
Presence of joint noises | Two months (every week with a total of six continuous records)
  Sound detected and recorded by the operator using a stethoscope placed in the anterior atrial area above the TMJ when making mandibular opening and closing movements.
Heart rate | Two months (every week with a total of six continuous records)
  Number of times the heart beats for one minute, measured with using a finger oximeter Pulox Oxímetro de Pulso PO-200. Number of beats Norm (60-100 beats)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Morales, Bachelor, Study Chair — Universidad Nacional Autonoma de Mexico

IPD SHARING:
Plan to Share IPD: Undecided
All collected IPD, all IPD that underlie results in a publication

REFERENCES:
- See also: Differences in masseter activity in patients with and without self-reported rheumatoid arthritis using surface electromyography: A cross-sectional study — https://www.researchgate.net/publication/334207017_Differences_in_masseter_activity_in_patients_with_and_without_self-reported_rheumatoid_arthritis_using_surface_electromyography_A_cross-sectional_study

DOCUMENTS (3):
  • Study Protocol (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04704778/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04704778/SAP_001.pdf
  • Informed Consent Form (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT04704778/ICF_002.pdf